CLINICAL TRIAL: NCT06439966
Title: Expanded Access to ABBV-787
Status: No longer available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C25-244
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: ABBV-787 — Intravenous (IV) Infusion

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to ABBV-787 prior to approval by the local regulatory agency. Availability will depend on territory eligibility. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Exclusion Criteria:

* There are other suitable treatment options.
* The participant qualifies for ongoing clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=C25-244